CLINICAL TRIAL: NCT05675150
Title: Unlocking Limitations Through Arts: A Mixed Methods Study on the Effectiveness of an Expressive Arts-based Intervention on Psychosocial Wellbeing of Adults With Age-related Visual Impairment
Brief Title: Expressive Arts-based Intervention for Adults With Age-related Visual Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Polytechnic University (Other); The Hong Kong Society for the Blind (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17611122
Record Dates: First submitted 2023-01-02; First posted 2023-01-09 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Age-Related Macular Degeneration
Keywords: Age-related visual impairment; Psychosocial wellbeing; Expressive arts-based intervention; Macular degeneration; Randomized controlled trial
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Intervention Model Description: Parallel Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of this trial, neither the staff, participants nor care provider can be masked to allocation. The data analyst will be blinded after study completion by having the intervention group information coded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This arm of participants will be receiving expressive arts-based intervention as intervention
  Interventions: Behavioral: Expressive Arts-Based Intervention
- Wait-list control (No Intervention): This arm of participants will not receive any art-based intervention during the study and are allocated as a wait-list control group

INTERVENTIONS:
Behavioral: Expressive Arts-Based Intervention — The intervention brings together the strengths of different art modalities, such as visual art, music, movement, dance, drama and writing to assist reflection and response in individuals to their personal issues. Such variety of art forms multiplies the avenues by which a person in intervention may seek meaning, clarity, insight and healing.
  Arms: Intervention

SUMMARY:
Age-related Macular Degeneration (AMD) is an age-related eye disease resulting in vision loss. Persons with AMD not only experience a gradual loss of ability in independent living, but also profound impairment in psychosocial well-being.The multimodal, expressive arts-based intervention (EXABI) that emphasizes imagination and creativity can be an engaging, enjoyable, and safe process of empowerment. This study aims to investigate the effectiveness and process of an expressive arts-based intervention in enhancing psychosocial wellness and adjustment to gradual vision loss of persons with AMD. This current study will adopt a 2-arm randomized controlled design with treatment-as-usual control. Upon screening for inclusion exclusion criteria, baseline data will be collected; and eligible participants will be randomized into either an 8-week Expressive Arts-based intervention group or Treatment-As-Usual control group.

DETAILED DESCRIPTION:
Age-related Macular Degeneration (AMD) is an age-related eye disease resulting in vision loss. Persons with AMD not only experience a gradual loss of ability in independent living, but also profound impairment in psychosocial well-being. Given the impacts of irreversible visual loss, persons with AMD need to actively adapt to changes and renegotiate supportive relations to maintain well-being. Psychosocial enhancement may buffer against the deteriorating quality of life, psychological distress, and poor adjustments among adults with AMD. The multimodal, expressive arts-based intervention (EXABI) that emphasizes imagination and creativity can be an engaging, enjoyable, and safe process of empowerment. The EXABI could help bypass or expand the limit of vision during interaction, and broaden the coping repertoire of those with AMD.

This study aims to investigate the effectiveness and process of an expressive arts-based intervention in enhancing psychosocial wellness and adjustment to gradual vision loss of persons with AMD. Primary outcomes include psychosocial adaptation, and vision-related quality of life; and secondary outcomes including symptoms of depression and anxiety, resilience, social support, and imagination as well as associations between psychosocial variables, participants' experience in the group, and factors affecting the effectiveness of the EXABI will be explored.

This proposed study adopts a randomized controlled trial with mixed methods design. To address the research objectives, data collected will be triangulated and interpreted simultaneously to address the research questions. Outcome measures will be assessed on four time-points (T0: Pre-intervention at baseline; T1: Post-intervention; T2: 3-month post-intervention and; T3: 6-month post-intervention) to assess the immediate and sustained effects of the expressive arts-based intervention on psychosocial wellbeing of the participants. Qualitative interviews will be conducted with a random subsample of 30 participants from the expressive arts group at T1 and T3 to collect fine-grained, information to explore their overall experience of participation in the intervention and how the experience has shaped their coping experience in terms of stress management, self-care challenges, and to reestablish severed social connections. Results of the qualitative interviews will be used to enhance the interpretation and understanding of the quantitative findings.

ELIGIBILITY:
Inclusion Criteria:

* Participants are community-dwelling, Chinese-speaking adults aged between 50 and 80, with the diagnosis of age-related macular degeneration in one or both eyes of all different etiologies

Exclusion Criteria:

* Inability to understand the Chinese language, as well as a diagnosis of total blindness, presence of other significant physical, psychological, and cognitive comorbidities that would hinder the participant from completing the study will be excluded.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Baseline Psychosocial Adaptation Questionnaire for visual impairment level at 2 months, 5 months, and 8 months | Baseline, post-intervention (Month 2), 3-month post-intervention (Month 5), and 6-month post-intervention (Month 8)
  Administration of the Chinese translated version of the 38-item Psychosocial Adaptation Questionnaire:
  * The first factor was attitude, involving 10 items. The second factor was self-acceptance, involving six items. The third factor was self-esteem involving six items. The fourth factor was anxiety/depression, involving six items. The fifth factor was belonging, involving five items. The sixth factor was self-efficacy involving three items. The last factor was the sense of self-control, involving two items.
  * Higher scores indicate a higher level of endorsement in a specific domain.
  * Likert's scale with four points was used to quantify results. The four points included completely incorrect, more correct, most correct, and completely correct. The score for positive items was one point, two points, three points, and four points; negative items were scored oppositely.
  * Q14, Q17, Q19, Q20, Q21, Q22, Q29, Q30, Q31, and Q32 are reversed (positive) items.
Change of Baseline Vision-related Quality of Life level at 2 months, 5 months, and 8 months | Baseline, post-intervention (Month 2), 3-month post-intervention (Month 5), and 6-month post-intervention (Month 8)
  Administration of the Chinese translated version of the 13-item Vision-related Quality of Life Scale:
  * Vision-specific quality of life is measured by the 13-item Vision-Related Quality of Life Scale taken from 25-item National Eye Institute Visual Function Questionnaire.
  * Social functioning of Vision-specific quality of life is Q11 and Q13 respectively.
  * Mental health of Vision-specific quality of life is Q3, Q25, Q21, and Q22 respectively.
  * Role limitation of Vision-specific quality of life is Q17 and Q18 respectively.
  * Dependency of Vision-specific quality of life is Q20, Q23, and Q24 respectively.
  * Ocular pain of Vision-specific quality of life is Q4 and Q19 respectively.
  * Original numeric values from the survey are re-coded following the scoring rules. All items are scored so that a high score represents better functioning. Each item is then converted to a 0 to 1

SECONDARY OUTCOMES:
Change of Baseline Anxiety level at 2 months, 5 months, and 8 months | Baseline, post-intervention (Month 2), 3-month post-intervention (Month 5), and 6-month post-intervention (Month 8)
  Administration of the Chinese translated version of the Hospital Anxiety and Depression Scale.
  * This scale is adopted to measure the level of Anxiety.
  * The minimum score is 0 and the maximum score is 21.
  * Scores ranging from "0-7" represents "Normal", ranging from "8-10" represents "Borderline abnormal", and ranging from "11-21" represents "Abnormal".
Change of Baseline Depression level at 2 months, 5 months, and 8 months | Baseline, post-intervention (Month 2), 3-month post-intervention (Month 5), and 6-month post-intervention (Month 8)
  Administration of the Chinese translated version of the Hospital Anxiety and Depression Scale.
  * This scale is adopted to measure the level of Depression.
  * The minimum score is 0 and the maximum score is 21.
  * Scores ranging from "0-7" represents "Normal", ranging from "8-10" represents "Borderline abnormal", and ranging from "11-21" represents "Abnormal".
Change of Baseline Resilience level at 2 months, 5 months and 8 months | Baseline, post-intervention (Month 2), 3-month after post-intervention (Month 5), and 6-month after post-intervention (Month 8)
  Administration of the Chinese translated version of the self-report Resilience Scale-14.
  * The brief "RS-14 scale consists of 14 self-report items measured along a 7-point rating scale ranging from '1-strongly disagree' to '7-strongly agree.'
  * Higher scores are indicative of resilience level.
  * Scores are calculated by a summation of response values for each item, thus enabling scores to range from 14 to 98.
  * Scores below 65 indicate low resilience; between 65 and 81 show moderate resilience; above 81 will be interpreted as high levels of resilience.
Change of Baseline Perceived Social Support level at 2 months, 5 months and 8 months | Baseline, post-intervention (Month 2), 3-month after post-intervention (Month 5), and 6-month after post-intervention (Month 8)
  Administration of the Chinese version of the Multidimensional Scale of Perceived Social Support
  * This scale has adopted the measure the level of perceived social support from family, friends, or significant other.
  * The mean score of perceived social support from "family" is calculated by summing across Q3, Q4, Q8, and Q11, then divide by 4 values.
  * The mean score of perceived social support from "friends" is calculated by summing across Q6, Q7, Q9, and Q12, then divide by 4 values.
  * The mean score of perceived social support from "significant other" is calculated by summing across Q1, Q2, Q5, and Q10, then divide by 4 values.
  * The mean total score is calculated by summing across all 12 items, then divide by 12 values.
  * The minimum mean score of each sub-score and the total score is 1 and the maximum mean score is 7.
Change of Baseline Imagination level at 2 months, 5 months, and 8 months | Baseline, post-intervention (Month 2), 3-month after post-intervention (Month 5), and 6-month after post-intervention (Month 8)
  Administration of the Chinese translated version of the Self-Descriptive Imagination questionnaire.
  * The Self-Descriptive Imagination Questionnaire consists of 25 items. Expressive imagination is Q4, Q5, Q12, Q7, and Q13 respectively. Openness to variations is Q16, Q19, Q17, and Q23 respectively. Instrumental imagination is Q8, Q11, and Q10 respectively. Past/future mindedness is Q2, and Q1 respectively. Conventionality is Q24 and Q25 respectively.
  * The questionnaires measured along a 7-point rating scale ranging from '1- strongly disagree' to '7-strongly agree.' Scores are calculated by a summation of response values for each item, Higher scores are indicative of imagination level.
Change of Baseline Imagination level at 2 months, 5 months, and 8 months | Baseline, post-intervention (Month 2), 3-month after post-intervention (Month 5), and 6-month after post-intervention (Month 8)
  Administration of the Chinese translated version of the Fantastic Reality Ability Measurement.
  * The Fantastic Reality Ability Measurement consists of 21 items. Coping is Q4, Q8, Q15, and Q20 respectively. Transcendence is Q17, Q10, Q21, Q12, Q18, and Q7 respectively. Playfulness is Q5, Q6, Q9, Q14, Q19, and Q2 respectively. Control is Q11, Q13, Q3, Q16, and Q1 respectively.
  * The questionnaires measured along a 7-point rating scale ranging from '1- strongly disagree' to '7-strongly agree.' Scores are calculated by a summation of response values for each item, Higher scores are indicative of imagination level.

CONTACTS AND LOCATIONS:
Overall Officials: Rainbow Ho, Principal Investigator — Director/Professor
Locations (1):
- Centre on Behavioral Health, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The data of this study are available from the principal investigator upon reasonable request. The data are not publicly available because they involve personal and clinical data from patients with age-related macular degeneration (AMD).
Supporting Information: Study Protocol, ICF
Time Frame: 3 years after the completion of the study
Access Criteria: The principal investigator will evaluate each request to determine if the data is accessible to other researchers.

REFERENCES:
- [Derived] Ho RTH, Cheong AMY, Wan AHY, Lo TLT, Fong TCT, Chan CKP, Li Q, Chan WC. Protocol for a mixed-methods randomised controlled trial evaluating the psychosocial effects of an expressive arts-based intervention on adults with age-related macular degeneration. BMJ Open. 2024 Dec 20;14(12):e088311. doi: 10.1136/bmjopen-2024-088311. PMID 39806623

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/50/NCT05675150/Prot_SAP_000.pdf